CLINICAL TRIAL: NCT01594138
Title: Linguistic Characteristics of Suicidal Patients in the ED (Emergency Department)
Brief Title: Linguistic Characteristics of Suicidal Patients in the Emergency Department
Status: Completed | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Other Study IDs: 2008-1421
Record Dates: First submitted 2012-04-30; First posted 2012-05-08 (Estimated); Last update posted 2017-02-15 (Actual); Status verified 2017-02

CONDITIONS: Suicide
MeSH Terms: conditions — Suicide

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Suicidal Subjects: Suicidal Subjects
  Interventions: Other: Standardized questionnaires and a ubiquitous questionnaire
- Non-Suicidal Control Subjects: Non-Suicidal Control Subjects
  Interventions: Other: Standardized questionnaires and a ubiquitous questionnaire

INTERVENTIONS:
Other: Standardized questionnaires and a ubiquitous questionnaire — Columbia Suicide Severity Rating Scale, Suicidal Ideation Questionnaire,Peabody Caregiver Background Form,CCHMC Suicide History Form,and ubiquitous questionnaire(UQ ver.2011)

SUMMARY:
The purpose of this study is to determine whether patients who have a high risk for serious suicide behavior will demonstrate a speech pattern that has a relationship to language patterns found in suicide notes.

DETAILED DESCRIPTION:
In an average week the CCHMC Emergency Department (ED) evaluates 40 patients with suicidal behavior. Currently, there is no systematic method for assessment of suicide risk in these patients and often, emergency department staff are required to make judgments about the disposition of these patients without a full understanding of the patient's risk for another serious suicide attempt. This pilot project involves experts in child psychiatry, biomedical informatics, and emergency medicine to collect pilot data for developing a method to estimate the risk of serious suicidal behavior based on computational linguistics.

ELIGIBILITY:
Inclusion Criteria for Suicidal Subjects:

* Subjects age 13 years 0 months to 17 years, 11 months old
* Admission to CCHMC ED, psychiatric units, or medical units with suicidal behavior or attempt
* The patient and legal guardian must understand the nature of the study and be able to comply with protocol requirements. The legal guardian must give written informed consent and the youth, written assent.
* English is spoken as the primary language in the home

Inclusion Criteria for Non-Suicidal Subjects:

* Subjects age 13 years 0 months to 17 years, 11 months old
* Admission to CCHMC ED with no current or no history of suicide ideation/attempt/gesture
* No past or current history of a major mood disorder
* No history of death by suicide in first-degree relatives
* The patient and legal guardian must understand the nature of the study and be able to comply with protocol requirements. The legal guardian must give written informed consent and the youth, written assent.
* English is spoken as the primary language in the home

Exclusion Criteria for Suicidal Subjects:

* Any serious, unstable medical illness or clinically significant abnormal laboratory assessments that would adversely impact the scientific interpretability or unduly increase the risks of the protocol
* Level of consciousness precludes consent and research assessments
* Unable to assent because of severe mental retardation or incapacitating psychosis

Exclusion Criteria for Non-Suicidal Subjects:

* Any current or past suicide attempts
* Any serious, unstable medical illness or clinically significant abnormal laboratory assessments that would adversely impact the scientific interpretability or unduly increase the risks of the protocol.

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: CCHMC suicidal and non-suicidal adolescents
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2009-09; Primary Completion 2011-11 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Differences between questionnaire responses from adolescents with and without suicidal behavior | At time of questinnaire administration

CONTACTS AND LOCATIONS:
Overall Officials: John Pestian, PhD, Principal Investigator — Cincinnati Childrens Hospital Medical Center
Locations (1):
- Cincinnati Children's Hopsital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available.